CLINICAL TRIAL: NCT06452043
Title: Nature-based Therapy Program for Sustainable Health in Parkinson's Disease (PARC Project) - a Clinical Trial
Brief Title: Nature-based Therapy Program for Parkinson's Disease (PARC)
Acronym: PARC
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Université du Québec à Chicoutimi (Other)
Collaborators: Réseau Parkinson Québec (Unknown); McGill University (Other); Fonds de la Recherche en Santé du Québec (Other Government)
Responsible Party: Principal Investigator, Rubens da Silva, Director and professor, Université du Québec à Chicoutimi
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 2024-1664
Record Dates: First submitted 2024-05-22; First posted 2024-06-11 (Actual); Last update posted 2024-12-06 (Actual); Status verified 2024-12

CONDITIONS: Chronic Disease; Fall Patients; Aging Problems; Parkinson Disease
Keywords: Aging; Rehabilitation; Postural control; Falls; Biomechanics; Well-being; Social; Mobility; Strength; Nature-based therapy; Shinrin-Yoku; Forest bathing; Mindfulness; Meditation; Physical activity
MeSH Terms: conditions — Chronic Disease; Parkinson Disease; Motor Activity

STUDY DESIGN:
Intervention Model Description: Clinical trial design
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (1):
- Nature-based intervention (Experimental): Nature-based group intervention of once a week for 8 weeks
  Interventions: Other: PARC program

INTERVENTIONS:
Other: PARC program — Activities in nature such as walking, exercises (strengthening, mobility, balance), pedal boat, yoga, dance, mindfulness, meditation, forest bathing or Shinrin-Yoku, interpretation of nature
  Other Names: Nature-based therapy

SUMMARY:
The goal of this clinical trial is to learn if a nature-based program has positive effects on the physical and psychosocial health in a group of participants with Parkinson's disease. The main questions it aims to answer are:

Will the program improve:

* The physical outcomes such as mobility, strength and balance?
* The psychosocial health outcomes?

Participants will:

* Be assessed before and after the program;
* Participate in one session per week of the intervention.

DETAILED DESCRIPTION:
The chronic and neurodegenerative disease of Parkinson's (PD) is often characterized by movement and balance disorders, which are accompanied by an increased risk of falls. Falls are one of the most common problems that can lead to subsequent injuries (e.g., femoral head fracture) and associated mortality rates. Falls are frequent, debilitating, and have deleterious effects on self-confidence and the quality of life of individuals with PD. Additionally, according to Parkinson Canada, a high proportion of individuals living with this disease suffer from depression and/or anxiety. Therefore, it is essential to implement intervention programs aimed at improving the physical and functional capacity as well as the well-being of this population to prevent falls and promote sustainable health.

In recent years, an increasing number of studies have demonstrated the benefits of contact with nature on the physical and mental health of individuals. Specific and positive effects on psychological symptoms (e.g., depression) as well as cognition (memory) in adults have also been shown according to this recent evidence. This stimulates our research team to test the effects of a physical intervention in nature on the physical and mental health of individuals suffering from PD. One of the perspectives of this new intervention in nature is also to evaluate its impact on fall risks in this population. The ultimate goal of this project is to contribute to the sustainable health of the population.

The overall objective of this project, based on a pilot study, is to assess the effects of an 8-week nature-based intervention program on the physical and mental health of individuals with PD. Various physical measures (mobility, strength, and balance) and mental measures (level of depression, stress) will be studied in this project to better understand the effects of this type of intervention.

ELIGIBILITY:
Inclusion Criteria:

* diagnosed with Parkinson's disease (while medicated: ON);
* capable of walking independently;
* presenting mild to moderate disability symptoms according to the Hoehn and Yahr scale (stages 1-3);
* having a frailty score of less than 2/5 (Fried);
* having a cognitive status ≥26 based on the Mini-Mental State Examination (MMSE) questionnaire.

Exclusion Criteria:

* Cancer;
* Red flags (infection, tumor, etc.);
* Severe psychiatric disorders;
* Palliative care;
* Severe systemic syndromes or diseases that may prevent tests and exercises from being performed;
* Stroke - very acute phase (1 week) and this until medial hemodynamic stability.

Ages: 45 Years to 85 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 11 (Actual)
Dates: Start 2024-08-05 (Actual); Primary Completion 2024-10-07 (Actual); Study Completion 2024-10-07 (Actual)

PRIMARY OUTCOMES:
Postural control | change from baseline at 0 to 8 weeks
  Measures of center of pressure (COP) from plateform of force during different balance tasks
Walking | change from baseline at 0 to 8 weeks
  Gait parameters from GaitRite measurement The participants will be asked to walk at normal and fast speeds on a GaitRite treadmill (GAI-TRite® Platinum) Plus System 16' - 4.876 m, SN: Q209, CIR Systems Inc., Franklin, NJ, USA). Participants will perform each task twice. Main gait parameters will be used as main outcomes such as velocity in m/s.
Well-being state (WHO-5) | change from baseline at 0 to 8 weeks
  The World Health Organization Well-Being Index (WHO-5) is a widely used self-reported questionnaire designed to measure subjective well-being. It assesses the individual's overall psychological well-being and quality of life. The WHO-5 consists of five simple questions that ask respondents to rate their well-being over the past two weeks. The questions cover aspects such as positive mood, vitality, and general interest in life.
  The questionnaire is scored on a scale from 0 to 100, with higher scores indicating better well-being.
Depression state (PHQ-9) | change from baseline at 0 to 8 weeks
  The Patient Health Questionnaire-9 (PHQ-9) is a self-administered tool used to screen, diagnose, monitor, and measure the severity of depression. It consists of nine questions based on the diagnostic criteria for major depressive disorder in the DSM-5 (Diagnostic and Statistical Manual of Mental Disorders, Fifth Edition).Respondents rate how often they have experienced each symptom over the past two weeks on a scale ranging from 0 (not at all) to 3 (nearly every day). The scores are then added together to produce a total score ranging from 0 to 27, with higher scores indicating greater severity of depressive symptoms
Social Provisions (SPS-10) | change from baseline at 0 to 8 weeks
  The Social Provisions Scale-10 (SPS-10) is a shorter version of the original Social Provisions Scale (SPS). It is a brief self-report questionnaire designed to measure perceived social support across five dimensions. The SPS-10 is derived from the longer SPS but consists of a subset of items that capture key aspects of social support.
  Similar to the original SPS, respondents rate their agreement with each item on a Likert scale, ranging from 1 (strongly disagree) to 4 (strongly agree). The SPS-10 provides a quick and efficient way to assess an individual's perceived social support network and their satisfaction with various aspects of their social relationships.
Connection to nature (CNS) | change from baseline at 0 to 8 weeks
  The Connection to Nature Scale (CNS) is a psychological assessment tool designed to measure an individual's subjective connection to nature. It evaluates the degree to which people perceive themselves as a part of the natural world and the extent to which they appreciate and value nature in their lives.
  Respondents are asked to rate their agreement with each statement on a Likert scale, ranging from 1 (strongly disagree) to 5 (strongly agree). The scores are then totaled to provide an overall measure of an individual's connection to nature.

SECONDARY OUTCOMES:
Functional mobility test (TUG) | change from baseline at 0 to 8 weeks
  To assess mobility. Equipment: A stopwatch. Directions: Patients wear their regular footwear and can use a walking aid, if needed. Begin by having the patient sit back in a standard arm chair and identify a line 3 meters, or 10 feet away, on the floor.
5 times Sit-To-Stand (FTSTS) | change from baseline at 0 to 8 weeks
  f the 30 second sit to stand test was not applied for some patients, we used also this test which it measures the amount of time it takes for a patient to sit and stand five times in succession with arms folded across their chest. 2 trials were applied in this test and the best time in seconds used for analysis.
Maximal isometric hand grip strength | change from baseline at 0 to 8 weeks
  Jamar dynamometer to assess maximal isometric hand grip strength and frailty criteria. 3 trials of maximal contraction up 5 seconds. The best value was retained and corrected by body mass index from Fried classification.
Number of falls | change from baseline at 0 to 8 weeks
  Self-reported falls before, during and after the study
Trunk postural control on wobble chair | change from baseline at 0 to 8 weeks
  This test measures trunk postural balance during a sitting balance task on an unstable chair where only lumbar spine movements are allowed to restore balance. Briefly, the base of the chair consists of a pivot at its center and four springs that can be arranged and fixed at a distance varying between 6.0 and 21 cm from the center, allowing the system's level of stability to be varied. The system allows only forward/backward and lateral tilting.

OTHER OUTCOMES:
Falls Efficacy Scale-International (FES-I) | change from baseline at 0 to 8 weeks
  The Falls Efficacy Scale-International (FES-I) is a short, easy to administer tool that measures the level of concern about falling during social and physical activities inside and outside the home whether or not the person actually does the activity. The level of concern is measured on a four point Likert scale (1=not at all concerned to 4=very concerned)
Frailty criteria from Fried | change from baseline at 0 to 8 weeks
  The presence of frailty criteria according to Fried was assessed with self-report questions and two physical tests from five characteristics : 1) Low physical activity (to capture history of sedentary behavior or activity: ex. Do you get any physical exercise for the sake of exercising? How often do you leave your house?); 2) fatigue (complaint of exhaustion with normal activity such as walking outside, climbing stairs: ex. I felt that everything I did was an effort in the last week?); 3) weight loss (unintentional weight loss 10 lbs. or more in past year or more than 5% in past year); 4) weakness (grip strength evaluated with manual dynamometer; in average <30 kg for men and <18 kg for women, but data is normalized by body mass index); 5) slowness or slow walking speed (usual gait speed over 4.57 meters (15 feet); ex. >6.5 seconds, dependent of height).
Hoehn and Yahr Scale | Only at baseline from Sample characterization when Parkinson was included
  It is a five-point scale used by doctors and researchers to rate the degree of disability and severity of symptoms caused by Parkinson's disease:
  Stage 1: Unilateral involvement only Stage 1.5: Unilateral and axial involvement Stage 2: Bilateral involvement without impairment of balance Stage 2.5: Mild bilateral disease with recovery on pull test Stage 3: Mild to moderate bilateral disease; some postural instability; physically independent Stage 4: Severe disability; still able to walk or stand unassisted Stage 5: Wheelchair bound or bedridden unless aided
Cognitive status | Only at baseline from Sample characterization
  Mini-mental state questionnaire (MMSE or Folstein), which is used for grading the cognitive state of patients in this study. It's assessing the attention and orientation, memory, registration, recall, calculation, language and ability to draw a complex polygon.
  It is ranged from 0 to 30, where 30 means no impairment.

CONTACTS AND LOCATIONS:
Overall Officials: Rubens da Silva, PhD, Principal Investigator — Université du Québec à Chicoutimi; Marie-Ève Langelier, MD, Study Chair — Université du Québec à Chicoutimi; Émilie Fortin, PT, Study Chair — Université du Québec à Chicoutimi; Mireille Cliche, SW, Study Chair — Université du Québec à Chicoutimi
Locations (1):
- Rubens da Silva, Saguenay, Quebec, Canada

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Shen X, Wong-Yu IS, Mak MK. Effects of Exercise on Falls, Balance, and Gait Ability in Parkinson's Disease: A Meta-analysis. Neurorehabil Neural Repair. 2016 Jul;30(6):512-27. doi: 10.1177/1545968315613447. Epub 2015 Oct 21. PMID 26493731
- [Background] Ray S, Agarwal P. Depression and Anxiety in Parkinson Disease. Clin Geriatr Med. 2020 Feb;36(1):93-104. doi: 10.1016/j.cger.2019.09.012. Epub 2019 Sep 10. PMID 31733705
- [Background] Lee I, Choi H, Bang KS, Kim S, Song M, Lee B. Effects of Forest Therapy on Depressive Symptoms among Adults: A Systematic Review. Int J Environ Res Public Health. 2017 Mar 20;14(3):321. doi: 10.3390/ijerph14030321. PMID 28335541
- [Background] Frumkin H, Bratman GN, Breslow SJ, Cochran B, Kahn PH Jr, Lawler JJ, Levin PS, Tandon PS, Varanasi U, Wolf KL, Wood SA. Nature Contact and Human Health: A Research Agenda. Environ Health Perspect. 2017 Jul 31;125(7):075001. doi: 10.1289/EHP1663. PMID 28796634
- [Background] Hvingelby VS, Glud AN, Sorensen JCH, Tai Y, Andersen ASM, Johnsen E, Moro E, Pavese N. Interventions to improve gait in Parkinson's disease: a systematic review of randomized controlled trials and network meta-analysis. J Neurol. 2022 Aug;269(8):4068-4079. doi: 10.1007/s00415-022-11091-1. Epub 2022 Apr 5. PMID 35378605
- [Background] Sherrington C, Tiedemann A. Physiotherapy in the prevention of falls in older people. J Physiother. 2015 Apr;61(2):54-60. doi: 10.1016/j.jphys.2015.02.011. Epub 2015 Mar 18. PMID 25797882
- [Background] Han JW, Choi H, Jeon YH, Yoon CH, Woo JM, Kim W. The Effects of Forest Therapy on Coping with Chronic Widespread Pain: Physiological and Psychological Differences between Participants in a Forest Therapy Program and a Control Group. Int J Environ Res Public Health. 2016 Feb 24;13(3):255. doi: 10.3390/ijerph13030255. PMID 26927141
- [Background] Doll R. Chronic and degenerative disease: major causes of morbidity and death. Am J Clin Nutr. 1995 Dec;62(6 Suppl):1301S-1305S. doi: 10.1093/ajcn/62.6.1301S. PMID 7495224
- [Background] Song C, Ikei H, Park BJ, Lee J, Kagawa T, Miyazaki Y. Psychological Benefits of Walking through Forest Areas. Int J Environ Res Public Health. 2018 Dec 10;15(12):2804. doi: 10.3390/ijerph15122804. PMID 30544682
- [Background] Dallaire M, Houde-Thibeault A, Bouchard-Tremblay J, Wotto EA, Cote S, Santos Oliveira C, Ngomo S, da Silva RA. Impact of frailty and sex-related differences on postural control and gait in older adults with Parkinson's Disease. Exp Gerontol. 2024 Feb;186:112360. doi: 10.1016/j.exger.2024.112360. Epub 2024 Jan 13. PMID 38215954
- [Background] Fried LP, Tangen CM, Walston J, Newman AB, Hirsch C, Gottdiener J, Seeman T, Tracy R, Kop WJ, Burke G, McBurnie MA; Cardiovascular Health Study Collaborative Research Group. Frailty in older adults: evidence for a phenotype. J Gerontol A Biol Sci Med Sci. 2001 Mar;56(3):M146-56. doi: 10.1093/gerona/56.3.m146. PMID 11253156
- [Background] Terra MB, Da Silva RA, Bueno MEB, Ferraz HB, Smaili SM. Center of pressure-based balance evaluation in individuals with Parkinson's disease: a reliability study. Physiother Theory Pract. 2020 Jul;36(7):826-833. doi: 10.1080/09593985.2018.1508261. Epub 2018 Aug 17. PMID 30118638